CLINICAL TRIAL: NCT02997501
Title: Detect EGFR T790M Mutation in ctDNA of Chinese Advanced/Metastatic NSCLC Patients by Cobas, Super-ARMS, Digital PCR and NGS and Evaluate Clinical Outcomes of T790M Mutation Positive Patients Who Had AZD9291 Monotherapy
Brief Title: T790M Plasma Testing Methodology Comparison and Clinical Validation
Acronym: ADELOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: TigerMed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5160C00042
Record Dates: First submitted 2016-12-09; First posted 2016-12-20 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD9291 (Experimental): Single arm of AZD9291, starting dose of 80mg
  Interventions: Procedure: T790M+ Testing; Procedure: Baseline Visit Blood & Urine Testing; Procedure: Baseline ECG; Procedure: Visual Slit-Lamp Testing; Drug: AZD9291 Dosing; Procedure: Plasma AZD9291 testing

INTERVENTIONS:
Procedure: T790M+ Testing — The patient will need to have T790M+ testing
Procedure: Baseline Visit Blood & Urine Testing — Blood count and standard chemistry testing to ensure patient meets inclusion/exclusion criteria
Procedure: Baseline ECG — ECG to ensure absence of any cardiac abnormality
Procedure: Visual Slit-Lamp Testing — Slit-lamp testing performed to ensure patients do not have any eye abnormalities or symptoms
Drug: AZD9291 Dosing — Patients to be provided with AZD9291 every 6 weeks (+/- 7 days)
Procedure: Plasma AZD9291 testing — The patient will need to have plasma AZD9291 testing before treatment

SUMMARY:
The aim of this study is to evaluate concordance of T790M mutation plasma testing between the Cobas test and each of other platforms: Super-ARMS, digital PCR or NGS. And to assess the efficacy of AZD9291 monotherapy by assessment of PFS in adult patients with advanced or metastatic NSCLC, who have received prior EGFR-tyrosine kinase inhibitor (TKI) therapy and are T790M mutation positive detected by any one of the four plasma testing platforms: Cobas/Super-ARMS/ digital PCR/NGS.

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to evaluate concordance of T790M mutation plasma testing between the Cobas test and each of other platforms: Super-ARMS, digital PCR or NGS. And to assess the efficacy of AZD9291 monotherapy by assessment of PFS in adult patients with advanced or metastatic NSCLC, who have received prior EGFR-tyrosine kinase inhibitor (TKI) therapy and are T790M mutation positive detected by any one of the four plasma testing platforms: Cobas/Super-ARMS/ digital PCR/NGS.

Study number of patients planned: Approximately 250 patients will be recruited in China.

Study Design: This is an open-label, multi-center testing and treatment study.

Target patient population: 250 locally advanced or metastatic EGFR mutation positive NSCLC patients with progression on a previous EGFR-TKI will be recruited.

Investigational product (IP), dosage, and mode of administration: AZD9291 is an oral, potent, selective, irreversible inhibitor of both EGFR-TKI sensitizing and resistance mutations in NSCLC with a significant selectivity margin over wild-type EGFR. AZD9291 will be administered orally as one 80 mg tablet once a day. All AEs/SAEs would be reported in ASTRIS main study and would not be reported repeatedly in current study.

Duration of IP administration: Patients may continue to receive AZD9291 as long as they continue to show clinical benefit, as judged by the investigator, and in the absence of discontinuation criteria. The study will be closed in a maximum period of 18 months after the last patient is enrolled. Contingencies will be made to ensure continued drug supply for patients who are still deriving benefit from AZD9291 at that time.

Study measures: Data collected will include patient demographics, smoking history, information needed to determine patient eligibility (including medical history, past and current disease characteristics, and tumor EGFR mutations status, T790M and sensitizing mutations status results and type of test performed), AZD9291 exposure, investigator-reported efficacy (including tumor response and disease progression), overall survival (OS).

Statistical methods: The concordance of T790M resistance mutation testing between the Cobas test and each of other platforms will be calculated. The sensitivity, specificity, PPV and NPV of each testing platform (Super-ARMS, digital PCR, and NGS) will be calculated with the Cobas test as the reference. The Kappa coefficient will be calculated to measure the agreement of T790M mutation testing between the Cobas test and each of other platforms. Descriptive statistics will be provided for all variables, as appropriate. Continuous variables will be summarized by the number of observations, mean, standard deviation, median, interquartile range (Q1, Q3), minimum, and maximum. Categorical variables will be summarized by frequency counts and percentages for each category. The 95% confidence interval (CI) will be calculated as appropriate. PFS and OS, respectively, will be summarized using Kaplan-Meier estimates of the median time to event (progression and death) and quartiles together with their 95% confidence intervals.The chi-square test will be used to compare the sensitivity, specificity, and concordance between any of the two platforms using Cobas as reference testing in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Adults (according to China regulations for age of majority)
3. Histological or cytological confirmed locally advanced NSCLC (stage IIIB) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy.
4. Patients who have progressed following prior therapy with an EGFR-TKI agent.

Exclusion Criteria:

1. Patients who disagree to participate this study.
2. Patients whose medical objection was recorded to use the existing data from medical practice for scientific research.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yilong WU, Principal Investigator — Guangdong General Hospita; Zhiyong LIANG, Principal Investigator — Peking Union Medical College Hospital
Locations (5):
- China (5):
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Wuhan
  - Research Site, Xi'an

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00042&attachmentIdentifier=00838057-bf4d-4a07-a48d-743b0f2b20d5&fileName=D5160C00042_CSP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00042&attachmentIdentifier=9e0016e3-e49b-4686-999d-b4a4e3ba74de&fileName=D5160C00042_SAP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00042&attachmentIdentifier=34d8d065-9a6f-4218-8fc1-539d1be96542&fileName=D5160C00042-ADELOS-CSR.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Provision of informed consent prior to any study specific procedures.
  2. Adults (according to China regulations for age of majority).
  3. Histological or cytological confirmed locally advanced NSCLC (stage IIIB) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy.
  4. Patients who have progressed following prior therapy with an EGFR-TKI agent.
Pre-assignment Details: subjects with T790M+ in plasma were treated by AZD9291 and included in as-treated analysis set
Groups:
- Experimental: Patients who have progressed on previous EGFR-TKI receiving AZD9291 80mg PO QD.
Period: Overall Study
Arm/Group | Experimental
Started (2016-12-27) | 256 (receiveing AZD9291.)
Completed (2017-09-30) | 256
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.54 (9.506)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160
  Male | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 256
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
enrollment number [Count of Participants; unit: Participants]
  Patients who have progressed following prior therapy with an EGFR-TKI agent. | 256

OUTCOME MEASURES:

1. Primary Outcome: Concordance
Description: To evaluate concordance of T790M plasma mutation testing between the Cobas test and each of other platforms: Super-ARMS, digital PCR or NGS.
Time Frame: Up to 6 months
Measure: Number; unit: percentage of aggrement
Arm/Group | Experimental
Number analyzed (Participants) | 256
percentage of aggrement
  For T790M, referred to Cobas, the concordance for Super-ARMS | 91.3
  For T790M, referred to Cobas, the concordance for 3D PCR | 66.8
  For T790M, referred to Cobas, the concordance for NGS | 82.7
  For T790M, referred to Cobas, the concordance for ddPCR | 86.1
  For T790M, referred to Super-ARMS, the concordance for 3D PCR | 71.0
  For T790M, referred to Super-ARMS, the concordance for NGS | 88.3
  For T790M, referred to Super-ARMS, the concordance for ddPCR | 88.1
  For T790M, referred to 3D PCR, the concordance for NGS | 76.5
  For T790M, referred to 3D PCR, the concordance for ddPCR | 72.2
  For T790M, referred to NGS, the concordance for ddPCR | 85.8

2. Primary Outcome: PFS Using Investigator Assessments According to RECIST v1.1
Description: To assess the efficacy of AZD9291 monotherapy by assessment of PFS in adult patients with advanced or metastatic NSCLC, who have received prior EGFR- TKI therapy and are T790M mutation positive detected by any one of the four plasma testing platforms. PFS was defined using Response Evaluation Criteria In Solid Tumors version 1.1(RECIST v1.1).
Time Frame: The time from first dose of AZD9291 in this study until the date of disease progression as recorded in CRF or death (by any cause in the absence of progression), assessed up to 18 months
Population: Analysis population included AS-treated Analysis Set which contains all T790M postive patients via at least one of platforms. Patients with T790M positive results tested by each platform were also analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 167
months
  As-treated Analysis Set (contained all patients who took at least one dose of AZD9291) | 9.7 [8.4 to 11.2]
  T790M Positive in Plasma via Cobas at Baseline: number analyzed (Participants) | 89
  T790M Positive in Plasma via Cobas at Baseline | 10.6 [8.5 to 13.8]
  T790M Positive in Plasma via Super-ARMS at Baseline: number analyzed (Participants) | 101
  T790M Positive in Plasma via Super-ARMS at Baseline | 10.6 [8.7 to 12.5]
  T790M Positive in Plasma via 3D PCR at Baseline: number analyzed (Participants) | 148
  T790M Positive in Plasma via 3D PCR at Baseline | 9.7 [8.3 to 11.3]
  T790M Positive in Plasma via NGS at Baseline: number analyzed (Participants) | 129
  T790M Positive in Plasma via NGS at Baseline | 11.0 [9.5 to 13.8]
  T790M Positive in Plasma via ddPCR at Baseline: number analyzed (Participants) | 110
  T790M Positive in Plasma via ddPCR at Baseline | 10.5 [8.3 to 12.7]

3. Secondary Outcome: Testing Sensitivity, Specificity, PPV, NPV
Description: To evaluate the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of Super-ARMS/digital PCR/NGS by using Cobas as the reference.
Time Frame: Up to 6 months.
Measure: Number; unit: percentage
Arm/Group | Experimental
Number analyzed (Participants) | 256
percentage
  sensitivity for Super-ARMS | 94.7
  sensitivity for 3D PCR | 90.5
  sensitivity for NGS | 98.9
  sensitivity for ddPCR | 98.9
  specificity for Super-ARMS | 89.3
  specificity for 3D PCR | 52.5
  specificity for NGS | 73.0
  specificity for ddPCR | 78.5
  PPV for Super-ARMS | 84.1
  PPV for 3D PCR | 53.4
  PPV for NGS | 68.6
  PPV for ddPCR | 73.0
  NPV for Super-ARMS | 96.6
  NPV for 3D PCR | 90.2
  NPV for NGS | 99.1
  NPV for ddPCR | 99.2

4. Secondary Outcome: Overall Response Rate (ORR)
Description: To assess the efficacy of AZD9291 monotherapy by assessment of ORR in adult patients who have received prior EGFR-TKI therapy and are EGFR T790M mutation positive detected by any one of the four plasma testing platforms. ORR is defined as the percentage of patients with measurable disease with at least 1 visit response of CR or PR. Data obtained until progression or last evaluable assessment in the absence of progression will be included in the assessment of ORR.
Time Frame: From first patient first CT scan for RECIST assessment, till the last patient last CT scan, up to 22 months.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 167
percentage of participants
  As-treated Analysis Set | 56.3 [48.4 to 63.9]
  T790M Positive in Plasma via Cobas at Baseline: number analyzed (Participants) | 89
  T790M Positive in Plasma via Cobas at Baseline | 60.7 [49.7 to 70.9]
  T790M Positive in Plasma via Super-ARMS at Baseline: number analyzed (Participants) | 101
  T790M Positive in Plasma via Super-ARMS at Baseline | 62.4 [52.2 to 71.8]
  T790M Positive in Plasma via 3D PCR at Baseline: number analyzed (Participants) | 148
  T790M Positive in Plasma via 3D PCR at Baseline | 54.1 [45.7 to 62.3]
  T790M Positive in Plasma via NGS at Baseline: number analyzed (Participants) | 129
  T790M Positive in Plasma via NGS at Baseline | 62.0 [53.1 to 70.4]
  T790M Positive in Plasma via ddPCR at Baseline: number analyzed (Participants) | 110
  T790M Positive in Plasma via ddPCR at Baseline | 59.1 [49.3 to 68.4]

5. Secondary Outcome: 75% OS Duration
Description: To assess the efficacy of AZD9291 monotherapy by assessment of overall survival (OS) in adult patients who have received prior EGFR-TKI therapy and are EGFR T790M mutation positive detected by any one of the four plasma testing platforms. 75% OS duration was calculated.
Time Frame: From first patient signed the consent to study completion, up to 22 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental
Number analyzed (Participants) | 167
months
  As-treated Analysis Set | 9.7 [7.5 to 12.7]
  T790M Positive in Plasma via Cobas at Baseline: number analyzed (Participants) | 89
  T790M Positive in Plasma via Cobas at Baseline | 10.5 [7.3 to 13.6]
  T790M Positive in Plasma via Super-ARMS at Baseline: number analyzed (Participants) | 101
  T790M Positive in Plasma via Super-ARMS at Baseline | 10.7 [8.0 to 14.5]
  T790M Positive in Plasma via 3D PCR at Baseline: number analyzed (Participants) | 148
  T790M Positive in Plasma via 3D PCR at Baseline | 8.7 [7.3 to 12.1]
  T790M Positive in Plasma via NGS at Baseline: number analyzed (Participants) | 129
  T790M Positive in Plasma via NGS at Baseline | 11.9 [8.7 to 15.3]
  T790M Positive in Plasma via ddPCR at Baseline: number analyzed (Participants) | 110
  T790M Positive in Plasma via ddPCR at Baseline | 10.6 [8.0 to 14.3]

ADVERSE EVENTS:
Description: The main purpose of this study was to compare testing performance of different blood testing platforms and their guidance values to AZD9291. So this study didn't collect any drug safety data. It can be referred in the study protocol (Part 5.2) which showed safety assessments was not applicable in this study.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT02997501/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT02997501/SAP_001.pdf